CLINICAL TRIAL: NCT03462524
Title: Neoadjuvant Therapy for Locally Advanced Esophageal Cancer: Impact on Cardiopulmonary Physiology, Short- and Long-term Morbidity
Brief Title: Neoadjuvant Therapy for Esophageal Cancer and Cardiopulmonary Physiology
Status: Completed | Type: Observational
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Surgical Research Fellow, St. James's Hospital, Ireland
Other Study IDs: SJHDOS201701
Record Dates: First submitted 2018-02-28; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Cancer; Radiation Pneumonitis; Pulmonary Fibrosis; Respiratory Failure; Pneumonia; Surgery; Chemotherapy Effect; Radiation Fibrosis; Radiation Toxicity; Adenocarcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Radiation Pneumonitis; Pulmonary Fibrosis; Respiratory Insufficiency; Pneumonia; Radiation Fibrosis Syndrome; Radiation Injuries; Adenocarcinoma; Carcinoma, Squamous Cell | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant chemotherapy
  Interventions: Procedure: Esophagectomy
- Neoadjuvant chemoradiation
  Interventions: Procedure: Esophagectomy

INTERVENTIONS:
Procedure: Esophagectomy — FEV1, FVC and DLCO will be assessed at baseline and one month post induction therapy. Radiation induced lung injury (RILI EORTC grade≥2), CCI, Clavien-Dindo, and pulmonary complications will be monitored. Changes in pulmonary function will be compared with cardiorespiratory symptoms and HR-QL among disease-free survivors.

SUMMARY:
Although recent global trends indicate reduced postoperative mortality after esophagectomy, major morbidity, in particular pulmonary, remains high, with considerable health and economic costs. In a recent modern international collaborative series of 2704 patients from high-volume centers, with an approximate equal mix of open and minimally invasive approaches, respiratory complications were evident in 28% of patients, pneumonia in 15%, and respiratory failure in 7%.1 In other series, respiratory failure is reported in up to 15% of patients and is the most common cause of mortality. Prediction of risk and prevention of respiratory morbidity is therefore of considerable importance, and in this context baseline assessment of respiratory physiology compliments clinical assessment, history and enhanced recovery pathways representing key elements of current patient management.

In this study, which will include all prospective patients with locally advanced esophageal cancer treated at a National Center, pulmonary function will be systematically measured before and after neoadjuvant therapy. The investigators seek to evaluate the incidence of radiation induced lung injury (RILI), as well as subclinical changes in pulmonary physiology that may be linked to postoperative complications, and quality-of-life in survivorship, and to compare cohorts who received radiation therapy or chemotherapy alone, preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced esophageal cancer undergoing multimodal therapy with curative intent at study centre during study period
* Pulmonary function assessed at a minimum of one preoperative timepoint

Exclusion Criteria:

* Salvage, palliative or emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Records for all patients with LAEC treated with multimodal therapy with curative intent between 2010 and 2016 will be assessed for inclusion. Patients undergoing emergent or palliative surgery, or salvage esophagectomy will be excluded. All eligible patients for whom pulmonary function testing was undertaken at our Centre at a minimum of one preoperative timepoint will be included for analysis of operative and/or oncologic outcome. Then, HR-QL among disease-free patients at least one year postoperatively will be assessed using validated questionnaires (EORTC QLQC30, OG25 and OES18).
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 following administration of neoadjuvant chemotherapy versus chemoradiation | 4-6 weeks post completion of neoadjuvant therapy
  Changes in FEV1 (forced expiratory volume in one second, litres), both as a raw value, and as percentage of predicted values normalized for ethnicity, sex, age and height according to Global Lung Function Initiative algorithms will be determined.
Change in FVC following administration of neoadjuvant chemotherapy versus chemoradiation | 4-6 weeks post completion of neoadjuvant therapy
  Changes in FVC (forced vital capacity, litres), both as a raw value, and as percentage of predicted values normalized for ethnicity, sex, age and height according to Global Lung Function Initiative algorithms will be determined.
Change in DLCO following administration of neoadjuvant chemotherapy versus chemoradiation | 4-6 weeks post completion of neoadjuvant therapy
  Changes in DLCO (pulmonary diffusion capacity for carbon monoxide, mmol·min.-1.kPa. -1), both as a raw value, and as percentage of predicted values normalized for ethnicity, sex, age and height according to Global Lung Function Initiative algorithms will be determined.
Incidence of postoperative pulmonary morbidity as per Esophagectomy Complications Consensus Group (ECCG) definitions | Up to 90 days postoperatively
  Incidence of postoperative pulmonary morbidity, defined according to ECCG guidelines, will be compared after neoadjuvant chemotherapy versus chemoradiation.
Global health-related quality of life (HR-QL) score as assessed by Eastern Co-operative Oncology Group QLQ-C30 questionnaire | One year postoperatively
  "Global health" HR-QL scores at one year postoperatively among disease-free patients will be compared between neoadjuvant chemotherapy and chemoradiation cohorts

SECONDARY OUTCOMES:
Disease-free survival | To date of study completion or date of disease recurrence, whichever occurs first, with a minimum of one year follow-up for all surviving patients
  Disease-free survival will be compared between neoadjuvant chemotherapy and chemoradiation groups using Kaplan-Meier methods, as well as multivariable Cox proportional hazards regression models adjusting for known prognostic factors.
Overall survival | To date of study completion or date of death, whichever occurs first, with a minimum of one year follow-up for all surviving patients
  Disease-free survival will be compared between neoadjuvant chemotherapy and chemoradiation groups using Kaplan-Meier methods, as well as multivariable Cox proportional hazards regression models adjusting for known prognostic factors.

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Department of Surgery, St. James's Hospital, Dublin
  - Wellcome Trust-Health Research Board Clinical Research Facility, St. James's Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Undecided